CLINICAL TRIAL: NCT02660281
Title: Haploidentical Donor Hematopoietic Stem Cell Transplantation
Brief Title: URMC Related Haplo-identical Donor BMT
Acronym: HaploOnly
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Jeffrey Andolina, Medical Director, Pediatric BMT, University of Rochester
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UBMT 15056
Record Dates: First submitted 2015-11-24; First posted 2016-01-21 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-11

CONDITIONS: Hematological Disease; Immune Deficiencies; Solid Tumors; Myelofibrosis; Multiple Myeloma; Lymphoma
MeSH Terms: conditions — Hematologic Diseases; Primary Myelofibrosis; Multiple Myeloma; Lymphoma | interventions — fludarabine; Busulfan; Melphalan; Thiotepa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Full Intensity TBI-based Conditioning (Other): Total Body Irradiation 1200 cGy of 150 cGy over 4 or 5 days, days -5 or -4 to -1 Fludarabine 30 mg/m2/day x 3 days, days -6, -5, -4 Stem Cell Infusion, day 0 Post- Stem Cell Infusion Cyclophosphamide 50 mg/kg/day x 2 days, days +3 and +4 Mesna 50 mg/kg/day x 2 days, days +3 and +4
  Interventions: Radiation: Total Body Irradiation 1200 cGy; Drug: Fludarabine; Procedure: Stem Cell Infusion; Drug: Post-Stem Cell Infusion Cyclophosphamide; Drug: Post-Stem Cell Infusion Mesna
- Full Intensity Chemo-Only Conditioning (Other): Fludarabine 25 mg/m2/day x 5 days, days -6, -5, -4, -3, -2 Busulfan 130 mg/m2/day x 4 days, days -6, -5, -4, -3 Pre-Stem Cell Infusion Cyclophosphamide 14.5 mg/kg/day x 2 days, days -3 and -2 Pre-Stem Cell Infusion Mesna 14.5 mg/kg/day x 2 days, days -3 and -2 Stem Cell Infusion, day 0 Post-Stem Cell Infusion Cyclophosphamide 50 mg/kg/day x 2 days, days +3 and +4 Post-Stem Cell Infusion Mesna 50 mg/kg/day x 2 days, days +3 and +4
  Interventions: Drug: Fludarabine; Drug: Pre-Stem Cell Infusion Cyclophosphamide; Drug: Pre-Stem Cell Infusion Mesna; Drug: Busulfan; Procedure: Stem Cell Infusion; Drug: Post-Stem Cell Infusion Cyclophosphamide; Drug: Post-Stem Cell Infusion Mesna
- Reduced Intensity Conditioning (Other): Fludarabine 30 mg/m2/day x 5 days, days -6 to -2 Melphalan 140 mg/m2/day x 1 day, day -2 Stem Cell Infusion, day 0 Post-Stem Cell Infusion Cyclophosphamide 50 mg/kg/day x 2 days, days +3 and +4 Post-Stem Cell InfusionMesna 50 mg/kg/day x 2 days, days +3 and +4
  Interventions: Drug: Fludarabine; Drug: Melphalan; Procedure: Stem Cell Infusion; Drug: Post-Stem Cell Infusion Cyclophosphamide; Drug: Post-Stem Cell Infusion Mesna
- Non-Myeloablative Conditioning (Other): Fludarabine 30 mg/m2/day x 5 days, days -6 to -2 Pre-Stem Cell Infusion Cyclophosphamide 14.5 mg/kg/day x 2 days, days -3 and -2 Pre-Stem Cell InfusionMesna 14.5 mg/kg/day x 2 days, days -3 and -2 Total Body Irradiation 200 cGy, day -1 Stem Cell Infusion, day 0 Post-Stem Cell Infusion Cyclophosphamide 50 mg/kg/day x 2 days, day +3 and +4 Post-Stem Cell Infusion Mesna 50 mg/kg/day x 2 days, day +3 and +4
  Interventions: Radiation: Total Body Irradiation 1200 cGy; Drug: Fludarabine; Drug: Pre-Stem Cell Infusion Cyclophosphamide; Drug: Pre-Stem Cell Infusion Mesna; Procedure: Stem Cell Infusion; Drug: Post-Stem Cell Infusion Cyclophosphamide; Drug: Post-Stem Cell Infusion Mesna
- Reduced Intensity Conditioning with Addition of Thiotepa (Other): Fludarabine 30 mg/m2/day x 5 days, days -6 to -2 Thiotepa 8 mg/kg, day -3 Melphalan 140 mg/m2/day x 1 day, day -2 Stem Cell Infusion, day 0 Post-Stem Cell Infusion Cyclophosphamide 50 mg/kg/day x 2 days, days +3 and +4 Post-Stem Cell InfusionMesna 50 mg/kg/day x 2 days, days +3 and +4
  Interventions: Drug: Fludarabine; Drug: Melphalan; Procedure: Stem Cell Infusion; Drug: Post-Stem Cell Infusion Cyclophosphamide; Drug: Post-Stem Cell Infusion Mesna; Drug: Thiotepa

INTERVENTIONS:
Radiation: Total Body Irradiation 1200 cGy — 1200 cGy TBI in 8 fractions
  Other Names: TBI
  Arms: Full Intensity TBI-based Conditioning; Non-Myeloablative Conditioning
Drug: Fludarabine — Fludarabine
Drug: Pre-Stem Cell Infusion Cyclophosphamide — Cyclophosphamide given prior to the stem cell infusion
  Arms: Full Intensity Chemo-Only Conditioning; Non-Myeloablative Conditioning
Drug: Pre-Stem Cell Infusion Mesna — Mesna given prior to the stem cell infusion
  Arms: Full Intensity Chemo-Only Conditioning; Non-Myeloablative Conditioning
Drug: Busulfan — Busulfan
  Arms: Full Intensity Chemo-Only Conditioning
Drug: Melphalan — Melphalan
  Arms: Reduced Intensity Conditioning; Reduced Intensity Conditioning with Addition of Thiotepa
Procedure: Stem Cell Infusion — Stem cell infusion
Drug: Post-Stem Cell Infusion Cyclophosphamide — Cyclophosphamide given after the stem cell infusion
Drug: Post-Stem Cell Infusion Mesna — Mesna given after the Stem Cell Infusion
Drug: Thiotepa — Thiotepa
  Arms: Reduced Intensity Conditioning with Addition of Thiotepa

SUMMARY:
This study will be a single-center treatment protocol, designed to validate the process of related donor haploidentical-SCT at the Wilmot Cancer Institute Blood and Marrow Transplant Unit.

DETAILED DESCRIPTION:
This study will be a single-center treatment protocol with five possible preparative regimens, designed to validate the process of related donor haploidentical-SCT at the Wilmot Cancer Institute Blood and Marrow Transplant Unit. Enrolled patients will receive chemotherapy +/- radiation as a pre-transplant conditioning regimen. Patients will then receive haploidentical stem cells, either bone marrow or mobilized peripheral blood, followed by GvHD prophylaxis that will include cyclophosphamide. Multiple data points will be collected prior to, during, and following transplantation to ensure safety of the process and to evaluate the stated objectives.

ELIGIBILITY:
Inclusion Criteria:

Patient Age:

* Pediatric (ages 6 months to 18 years)
* Adult (ages 18-75 years)

Disease:

Congenital and Other Non-malignant Disorders

* Immunodeficiency disorders (e.g. Severe Combined Immunodeficiency, Wiskott-Aldrich Syndrome)
* Congenital hematopoietic stem cell defects (e.g. Chediak-Higashi Syndrome, Congenital Osteopetrosis, Osteogenesis Imperfecta)
* Metabolic disorders (e.g. Hurler's Syndrome)
* Hemoglobinopathies (e.g. Sickle Cell Disease, Thalassemia)
* Severe aplastic anemia

High-Risk Leukemias

Acute Myelogenous Leukemia

* Refractory to standard induction therapy (more than 1 cycle required to achieve remission)
* Recurrent (in CR≥2)
* Treatment-related AML or MDS
* Evolved from myelodysplastic syndrome
* Presence of Flt3 abnormalities
* FAB M6 or M7
* Adverse cytogenetics

Myelodysplastic Syndrome

Acute Lymphoblastic Leukemia including T lymphoblastic leukemia

* Refractory to standard induction therapy (time to CR >4 weeks)
* Recurrent (in CR ≥2)
* WBC count >30,000/mcL at diagnosis
* Age >30 at diagnosis
* Adverse cytogenetics, such as (t(9:22), t(1:19), t(4:11), other MLL rearrangements.

Chronic Myelogenous Leukemia in accelerated phase or blast crisis

Biphenotypic or undifferentiated leukemia

Burkitt's leukemia or lymphoma

Lymphoma:

* Large cell, Mantle cell, Hodgkin lymphoma refractory or recurrent, chemosensitive, and ineligible for an autologous stem cell transplant or previously treated with autologous SCT
* Marginal zone or follicular lymphoma that is progressive after at least two prior therapies

Multiple Myeloma, recurrent following high-dose therapy and autologous SCT or ineligible for an autologous HSCT

Solid tumors, with efficacy of allogeneic HSCT demonstrated for the specific disease and disease status

Graft failure following prior related donor, unrelated donor or UCB transplant

Myelofibrosis

Exclusion Criteria:

1. Patient Age below 6 months or over 75 years
2. Availability of a 10/10 HLA-matched related or unrelated donor within a reasonable time-frame dictated by the clinical urgency of the transplant
3. Autologous HSCT < 6 months prior to proposed haplo-SCT
4. Pregnant or breast-feeding
5. Current uncontrolled infection
6. Evidence of HIV infection or positive HIV serology
7. Anti-donor HLA antibodies with positive crossmatch and unsuccessful -

Ages: 6 Months to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2015-10; Primary Completion 2019-10-28 (Actual); Study Completion 2021-01-07 (Actual)

PRIMARY OUTCOMES:
The number of days from the date of the stem cell infusion to engraftment of absolute neutrophils (ANC) and platelets (PLT) will be determined based on daily CBC and differential counts. | 42 days following the infusion of stem cells for ANC. [If engraftment of ANC does not occur within 42 days, a subsequent transplant will be performed if a donor is available.
  The date of engraftment of ANC is the first of 3 consecutive days of ANC of 500 or higher. The date of engraftment of platelets is the first of 3 consecutive days of platelet counts of 20,000 or higher in the absence of platelet transfusions for at least 7 days prior.
Rate of non-engraftment and secondary graft failure | At 100 days, 6 months, and yearly after transplant from the date of transplant until the date of documented graft failure or the subject's date of death up to 120 months.
  The percentage of patients who fail to engraft ANC will be tabulated as well as the percentage of patients who have primary engraftment of ANC but whose graft then fails as evidenced by pancytopenia and failure of bone marrow function.

SECONDARY OUTCOMES:
Percentage of subjects who develop acute graft-versus-host disease. | 100 days following the infusion of stem cells
  Assess the presence and date of onset of acute GvHD based on the criteria published by Przepiorka et al., Bone Marrow Transplant 1995; 15(6):825-8 as used by the Center for International Blood & Marrow Transplant Research.
Assess the Maximum Overall Grades 0- IV of acute GvHD and Maximum Severity (0-4) by involved organ system in patients who develop acute graft-versus-host disease. | 100 days following the infusion of stem cells
  Assess the severity of acute GvHD based on the criteria published by Przepiorka et al., Bone Marrow Transplant 1995; 15(6):825-8 as used by the Center for International Blood & Marrow Transplant Research.
Percentage of subjects who develop chronic graft-versus-host disease. | Minimally at intervals of 100 days, 6 months and then yearly following the infusion of stem cells until the subject's date of death.or up to 120 months.
  Calculate the percentage of patients who develop chronic graft-versus-host disease based on Sullivan KM, Blood 1981; 57:267 as used by the Center for International Blood & Marrow Transplant Research.
Assess the Maximum Grade: Limited versus Extensive; Maximum Severity: Mild, Moderate or Severe) of chronic GvHD in patients who develop chronic graft-versus- | Minimally at intervals of 100 days, 6 months and then yearly following the infusion of stem cells until the subject's date of death or up to 120 months.
  Assess the severity of chronic GvHD in patients who develop chronic graft-versus-host disease based on Sullivan KM, Blood 1981; 57:267 as used by the Center for International Blood & Marrow Transplant Research.
Disease-free survival | Disease assessments are performed and reported at time points that include 100 days, 6 months, and yearly until documented progression of disease or the date of death or up to 120 months.
  Document and update the length of time a subject survives without recurrence of the disease for which they were transplanted minimally at 100 days. 6 months, and yearly following the infusion of stem cells for as long as the patient survives and remains disease-free.
Time to relapsed disease | Disease assessments are performed and reported at time points that include 100 days, 6 months, and yearly until the date of documented progression or the subject's date of death or up to 120 months.
  Document the time to relapse of the disease for which the patient was Minimally assessments will be performed at 100 days. 6 months, and yearly following the infusion of stem cells for as long as the patient survives and remains disease-free.
Immune reconstitution | At 100 day, 6 month and one year intervals following the infusion of stem cells until the subject's date of death or up to 120 months.
  Evaluate immune reconstitution by measurement of immunoglobulins (IgG, IgA, and IgM), assessment of infections, and lymphocyte analysis

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Andolina, MD, Principal Investigator — Wilmot Cancer Center
Locations (1):
- Wilmot Cancer Institute, Rochester, New York, United States